CLINICAL TRIAL: NCT07053644
Title: Community-derived Multilevel-Multicomponent Nutrition Intervention to Reduce Food Access Disparities -FRESH-EATS
Brief Title: FRESH-EATS Project
Acronym: FRESH-EATS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Heewon Gray, Associate Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY007833; R21MD019963 (NIH)
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Dietary Behaviors; Obesity and Overweight
Keywords: food insecurity; community-based; obesity prevention; nutrition education; behavioral intervention
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Research assistants who collect outcome data are blinded from the study condition. Study participants are also masked regarding their intervention condition when they participate in baseline data collection while they would naturally identify which condition they are in at the post-intervention assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants will receive multilevel multicomponent intervention FRESH-EATS. Four components include (1) Cooking lessons; (2) Family workshops addressing access to food; (3) Garden activities/education; and (4) Grocery delivery budget
  Interventions: Behavioral: FRESH-EATS
- Control (Active Comparator): Participants in the active comparison group will receive a six week education-only control intervention. After completing the post-intervention assessments, these families will receive the other components (family workshops, food delivery budget, and community garden involvement).
  Interventions: Behavioral: Lagged Intervention Control Group

INTERVENTIONS:
Behavioral: FRESH-EATS — 1. Six weekly Cooking Matters® for Families sessions. Each session is designed to take 90 minutes including hands-on cooking or other activities.
  2. Two 90-minute family workshop sessions will be implemented.
  3. Food delivery budget (i.e., the Walmart+ annual membership with free shipping and gift cards to purchase ingredients) will be provided up during the intervention period and local food pantry information will be distributed to families.
  4. Community garden at the Cornerstone Family Ministries will be utilized by incorporating garden activities, harvesting, and cooking with the produce from the garden.
  Arms: Intervention
Behavioral: Lagged Intervention Control Group — Nutrition education materials that address nutrition in school-age children and families Cooking Matters® for Families will be implemented. Each of six sessions will take about 90 minutes. All lessons will be delivered by qualified nutrition educators along with student assistants at the Cornerstone Family Ministries classrooms. After completing the post-intervention assessment, participants will then receive the other FRESH-EATS intervention components.
  Arms: Control

SUMMARY:
The goal of this randomized controlled trial is to determine the feasibility of the FRESH-EATS project in children ages 8-12 and their parents/caregivers residing in low-income, predominantly minority neighborhoods. The main questions it aims to answer are:

Is the FRESH-EATS intervention feasible to implement and well-received by parent-child dyads? Does the FRESH-EATS multilevel multicomponent intervention improve dietary behaviors of children and their parents/caregivers compared to the comparison group?

We hypothesize that this innovative community-derived, multilevel-multicomponent intervention is feasible to implement and has the potential to improve dietary behaviors of participants (children ages 8-12 and their parents/caregivers).

Researchers will compare the FRESH-EATS intervention group to the Lagged Intervention Control Group (LICG) to see if the FRESH-EATS intervention leads to better dietary behaviors and health outcomes.

Participants in the FRESH-EATS intervention group will:

* Attend educational sessions on healthy eating and cooking.
* Participate in family workshops that address access to healthy food.
* Receive food deliveries and information about local food resources.
* Engage in community garden activities.

DETAILED DESCRIPTION:
The FRESH-EATS project is a comprehensive intervention designed to address food access disparities and improve dietary behaviors among families in low-income neighborhoods. The intervention includes four key components. This program is tailored for school-aged children (ages 8-12) and their parents/caregivers, focusing on healthy eating as a family. Eight cohorts, each consisting of 6 families (48 families in total), will be recruited. Four cohorts (24 families) will participate in the FRESH-EATS intervention, while the other four cohorts (24 families) will be randomly assigned to the Lagged Intervention Control (LICG). The randomized controlled trial (RCT) design will compare the outcomes of the FRESH-EATS intervention group to the LICG group, with outcome evaluations conducted at both pre- and post-intervention stages.

First, it features evidence-based hands-on cooking and nutrition education using the Cooking Matters® for Families program. Additionally, the project includes family workshops aimed at addressing the lack of access to healthy foods and systemic disparities in the food environment. Throughout the intervention period, participants in the intervention group will receive food deliveries and information about local food resources such as food pantries. An updated list of local food pantries will be obtained from the local food bank. Handouts featuring different food pantries will be created and distributed to families. Intervention participants will receive community garden education that will provide fresh ingredients for participants to use during cooking lessons. The lead community organization has a community garden with 12 garden beds, which is active year-round in Florida. Season-specific garden education and activities will be integrated into the nutrition lessons, further supporting the project's goals of improving dietary behaviors and addressing food access disparities.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* Parents/caregivers that are 18 years or older
* Residents of targeted neighborhood
* Have a child aged 8-12 years old

Exclusion Criteria:

* Parents/caregivers or children who have participated in a similar intervention within the past 6 months
* Do not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Parent dietary behaviors | At baseline (T1) and post-intervention (T2) approximately 6-8 weeks from baseline.
  The Cooking Matters for Families Survey consists of 39 item, including questions on participants' dietary habits, meal preparation practices, food security, and attitudes towards healthy eating.
Children's dietary behaviors | At baseline (T1) and post-intervention (T2) approximately 6-8 weeks from baseline.
  Consists of 31 items. It assesses dietary intake of children including fruits, vegetables, beverages, and snack foods. The questionnaire is used to measure changes in these areas before and after an intervention

SECONDARY OUTCOMES:
Anthropometrics: height, weight, waist/hip circumferences | At baseline (T1) and post-intervention (T2) approximately 6-8 weeks from baseline.
  Assess children's height and weight with a professional stadiometer (SECA 213) and a weight scale (Tanita WB-800S) following the standardized protocol used in previous studies. As a standard weight status assessment for children, BMI percentile and z-scores based on the CDC growth chart will be calculated. Parent/caregiver BMI (kg/m²) will be calculated from waist and hip circumferences measurements collected by trained RAs using a circumference measuring tape (SECA 203).
Social Connectedness Scale | At baseline (T1) and post-intervention (T2) approximately 6-8 weeks from baseline.
  Scale consists of 20 items. It measures the extent to which individuals feel connected to others in their social environment, assessing dimensions such as belongingness, closeness, support, and satisfaction with social relationships. Each item is rated on a 6-point Likert scale, ranging from 1 (strongly disagree) to 6 (strongly agree)
Resilience | At baseline (T1) and post-intervention (T2) approximately 6-8 weeks from baseline.
  Connor-Davidson Resilience Scale consists of 10 items. It measures resilience, or the ability to cope with and bounce back from adversity. Each item is rated on a 5-point Likert scale, ranging from 0 (not true at all) to 4 (true nearly all the time). The total score ranges from 0 to 40, with higher scores indicating greater resilience.
Childhood Experiences Survey | At baseline (T1)
  An expanded and modified adverse childhood experiences assessment which consists of 17 questions including 10 conventional ACEs and 7 additional questions on financial problems, food insecurity, homelessness, death of a family member, prolonged parental absence, peer victimization, and violent crime victimization
Philadelphia Community- Level Adversity scale | At baseline (T1)
  This scale consists of 5 items. It measures community-level adversities such as witnessing violence, experiencing discrimination, living in an unsafe neighborhood, being bullied, and living in foster care. Each item is rated on a scale that reflects the frequency or intensity of these experience.
Perceived Food Access | At baseline (T1)
  Perceived food access data will be collected using six questions on perceptions of the food environment (e.g., how much of a problem would you say that lack of access to adequate food shopping is in your neighborhood?). The validity and reliability of these questions has been assessed in previous studies showing that the questions are valid and have good internal and test-retest reliability.
Blood Pressure | At baseline (T1) and post-intervention (T2) approximately 6-8 weeks from baseline.
  Parents/caregivers' and children's blood pressure will be measured with a digital monitor (CONTEC 08A) by trained RAs.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

REFERENCES:
- [Background] Gray HL, Berumen JH, Lovett SM, Himmelgreen D, Biswas D, Bohn J, Peacock C, Buro AW. A Mixed-methods Study to Understand Food Environments and Grocery Shopping Patterns of Community Residents in Underserved Neighborhoods in Tampa, Florida. Ecol Food Nutr. 2021 Jul-Aug;60(4):435-453. doi: 10.1080/03670244.2020.1862098. Epub 2020 Dec 23. PMID 33356564
- [Background] Hernandez DC, Reesor LM, Murillo R. Food insecurity and adult overweight/obesity: Gender and race/ethnic disparities. Appetite. 2017 Oct 1;117:373-378. doi: 10.1016/j.appet.2017.07.010. Epub 2017 Jul 22. PMID 28739148
- [Background] Reedy J, Krebs-Smith SM. Dietary sources of energy, solid fats, and added sugars among children and adolescents in the United States. J Am Diet Assoc. 2010 Oct;110(10):1477-84. doi: 10.1016/j.jada.2010.07.010. PMID 20869486
- [Background] Ghosh-Dastidar M, Hunter G, Collins RL, Zenk SN, Cummins S, Beckman R, Nugroho AK, Sloan JC, Wagner L, Dubowitz T. Does opening a supermarket in a food desert change the food environment? Health Place. 2017 Jul;46:249-256. doi: 10.1016/j.healthplace.2017.06.002. Epub 2017 Jun 22. PMID 28648926
- [Background] Chen D, Jaenicke EC, Volpe RJ. Food Environments and Obesity: Household Diet Expenditure Versus Food Deserts. Am J Public Health. 2016 May;106(5):881-8. doi: 10.2105/AJPH.2016.303048. Epub 2016 Mar 17. PMID 26985622
- [Background] Brown AG, Hudson LB, Chui K, Metayer N, Lebron-Torres N, Seguin RA, Folta SC. Improving heart health among Black/African American women using civic engagement: a pilot study. BMC Public Health. 2017 Jan 24;17(1):112. doi: 10.1186/s12889-016-3964-2. PMID 28118823
- [Background] Sankofa J, Johnson-Taylor WL. News coverage of diet-related health disparities experienced by black Americans: a steady diet of misinformation. J Nutr Educ Behav. 2007 Mar-Apr;39(2 Suppl):S41-4. doi: 10.1016/j.jneb.2006.08.014. PMID 17336804
- [Background] Larson NI, Story MT, Nelson MC. Neighborhood environments: disparities in access to healthy foods in the U.S. Am J Prev Med. 2009 Jan;36(1):74-81. doi: 10.1016/j.amepre.2008.09.025. Epub 2008 Nov 1. PMID 18977112
- [Background] Zenk SN, Odoms-Young AM, Dallas C, Hardy E, Watkins A, Hoskins-Wroten J, Holland L. "You have to hunt for the fruits, the vegetables": environmental barriers and adaptive strategies to acquire food in a low-income African American neighborhood. Health Educ Behav. 2011 Jun;38(3):282-92. doi: 10.1177/1090198110372877. Epub 2011 Apr 21. PMID 21511955
- [Background] Cubbin C, Hadden WC, Winkleby MA. Neighborhood context and cardiovascular disease risk factors: the contribution of material deprivation. Ethn Dis. 2001 Fall;11(4):687-700. PMID 11763293